CLINICAL TRIAL: NCT03016286
Title: Effects of Cooling of Ankle on Bone Myoregulation Reflex Response and Presynaptic Ia Inhibition Level
Brief Title: Bone Myoregulation Reflex & Presynaptic Ia Inhibition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, Head of PMR clinic, Bagcilar Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BMR20171
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Effects of Vibration
Keywords: Whole body vibration; Bone myoregulation reflex; H-reflex
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WBV group (Experimental): whole-body vibration (WBV) group
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — Whole body vibration at 25Hz frequency
  Other Names: Whole body vibration

SUMMARY:
Hypotheses of this study are

1. Bone myoregulation reflex (BMR) inhibits presynaptically H-reflex during whole-body vibration (WBV)
2. Cooling of ankle abolishes the inhibitor effect of BMR on soleus H-reflex Aim of this study is to test these hypotheses.

Methods: This study will be conducted on 10 healthy young adult males. WBV will be applied at 35 Hz frequencies with 2 mm amplitudes. Cold pack will be applied the right ankle for 20 minutes. The right soleus T-reflex will be recorded before WBV, during WBV, during cooling of the right ankle, and during WBV respectively.

DETAILED DESCRIPTION:
Hypotheses of this study are

1. Bone myoregulation reflex (BMR) inhibits presynaptically T-reflex during whole-body vibration (WBV)
2. Cooling of ankle abolishes the inhibitor effect of BMR on soleus T-reflex Aim of this study is to test these hypotheses.

Methods:

Participants:

Ten young, healthy and right hand dominant male adult volunteers will be included in this study.

Procedure:

Prior to the induction of WBV, control T-reflex recordings will be elicited and then the participants will complete a 15-s trial WBV protocol to familiarize themselves with the procedure. Following the control T-reflex recordings, the trial protocol and a 15-s rest, the participants will receive one session WBV. T-reflex will be recorded during WBV. Then, cold pack will be applied to the right ankle for 20 minutes. T-reflex will be recorded during the cooling of the ankle. Then, the participants will receive one session WBV, again. T-reflex will be recorded during WBV.

A light (2.9 gr.) triaxial (x, y and z-axis) accelerometer (LIS344ALH, ECOPACK®) will be taped on the right Achilles tendon so that the z-axis will be perpendicular with the direction of the tendon (Achilles accelerometer). A custom-made reflex hammer will be used to tap the right Achilles tendon just caudal to the accelerometer. The intensity of tapping will be about 19.6 N WBV frequencies of 35 Hz will be delivered for 60 s. The vibration plate of WBV device (Power-Plate®Pro5, PowerPlate® International, Ltd. London, UK) oscillates with a linear movement upward and downward. The participants will be barefooted and stand directly on the vibration platform. The surface electromyography (SEMG) data will be obtained while the participants stand upright on the vibration platform with the knees in extension. The Ag/AgCl electrodes (KENDALL®Covidien) with a disc radius of 10 mm will be placed 20 mm apart on the right soleus muscle belly on shaved skin in accordance with the recommendations of the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) project .

The recordings of both T-reflex and WBV-IMR will be acquired using SEMG. SEMG data will be recorded using a PowerLAB® data acquisition system (ADInstruments, Oxford, United Kingdom) and the data will be analyzed offline using the LabChart7® (ver 7.3.7, ADInstruments, Oxford, United Kingdom) software.

Precautions for voluntary muscle contractions and motion artifacts:

1. the participants will be asked to use the handles of the WBV device to secure their balance. The sense of balance may impair during WBV. Therefore muscles may be activated to restore balance during WBV,
2. before WBV trials, participants will be asked to relax and not to make voluntary contractions in their lower extremity muscles.
3. a trial protocol will be applied to familiarize vibration,
4. all cables will be carefully taped to the skin to minimize motion artifacts,
5. all EMG recordings will be filtered to avoid WBV induced movement artifacts using a band pass filter from 60 to 500 Hz.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Right-handed men

Exclusion Criteria:

* Bone, muscle/tendon, joint, vascular, dermatologic diseases in lower extremities and spine
* Medication that could affect the musculoskeletal system
* Postural abnormalities (scoliosis, kyphosis, etc)
* Systemic diseases

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-04-17 (Estimated); Study Completion 2018-04-17 (Estimated)

PRIMARY OUTCOMES:
Presynaptic Ia inhibition level | 1 month

IPD SHARING:
Plan to Share IPD: No